CLINICAL TRIAL: NCT01773759
Title: Strategies to Improve Vaccination Coverage in Child Care Centers and Preschools
Brief Title: Immunization Protection in Child Care (IPiCC) Project
Acronym: IPiCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Utah Department of Health (Other)
Responsible Party: Principal Investigator, Julie Shakib, Julie H. Shakib, DO, MPH, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IP000500; RFA-IP-11-006 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2013-01-13; First posted 2013-01-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Up-to-date Immunization Status for Children in Child Care
Keywords: Immunizations; Child care; School health promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention child care programs (Experimental): Intervention child care programs will receive immunization outreach and education.
  Interventions: Behavioral: Intervention child care programs
- Control child care programs (No Intervention): Control programs will receive no more than usual training regarding childhood immunization requirements.

INTERVENTIONS:
Behavioral: Intervention child care programs — Interventions will be designed based on findings from Aims 1 and 2, will include outreach and education, and may include on-site demonstration and USIIS training or peer tutoring.
  Arms: Intervention child care programs

SUMMARY:
Ensuring that all children are fully immunized against vaccine-preventable diseases is a critical public health issue. Child care programs are critical targets for efforts to increase the proportion of infants and young children who are fully immunized. The primary objective of this proposal is to rigorously examine current state, local government, and child care providers' efforts and barriers to ensuring that all enrolled children are up-to-date for required immunizations and to evaluate strategies to improve immunization coverage in child care programs.

DETAILED DESCRIPTION:
Specific Aim 1 will describe Utah state and local government activities to ensure compliance of child care programs with state immunization requirements and identify government's barriers to ensuring compliance.

Specific Aim 2 will describe child care program staffs' knowledge, attitudes, and activities related to ensuring that all children are up-to-date for required immunizations and identify program barriers to ensuring up-to-date status.

Specific Aim 3 will evaluate at least 3 strategies to ensure that all children enrolled in child care programs are up-to-date for required immunizations. Aims 1 and 2 will guide the design of these strategies. Specific strategies proposed for Aim 3 are to: 1) design and pilot test an intervention to increase child care program use of the Utah State Immunization Information System (USIIS), 2) design an online immunization education module and conduct a pilot randomized controlled trial to determine whether use of the module changes child care providers' knowledge, attitudes, and activities and increases the proportion of children who are up-to-date for required immunizations; and 3) conduct a pilot randomized controlled trial to determine whether a quality improvement intervention implemented in child care programs increases the proportion of children who are up-to-date for required immunizations.

ELIGIBILITY:
Inclusion Criteria:

Child care programs not currently registered to use the Utah State Immunization Information System (USIIS) in Utah counties with acceptable USIIS coverage will be included.

Exclusion Criteria:

Child care programs in Utah counties with lower than acceptable USIIS coverage will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Children enrolled in child care program up-to-date for required immunizations | Up to 2 years
  Proportion of children up-to-date for all state required childhood immunizations in the Utah State Immunization Information System (USIIS)

CONTACTS AND LOCATIONS:
Overall Officials: Julie H. Shakib, DO, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States